A Randomized Controlled Trial Comparing the Effect of Topical Dorzolamide-Timolol versus Placebo Combined with Intravitreal Anti-Vascular Endothelial Growth Factor (VEGF) Injections in Patients with Neovascular Age-Related Macular Degeneration Who Are Incomplete Anti-VEGF Responders

NCT03034772

**Document Date: 5/30/17** (statistical analysis finalized 2/4/20)

A Randomized Controlled Trial Comparing the Effect of Topical DorzolamideTimolol versus Placebo Combined with Intravitreal Anti-Vascular Endothelial

Growth Factor (VEGF) Injections in Patients with Neovascular Age-Related Macular Degeneration Who Are Incomplete Anti-VEGF Responders Principal Investigator: Jason Hsu, MD<sup>1</sup>

**Sub-investigators**: Chirag Shah, MD MPH<sup>2</sup>; Andre Witkin, MD<sup>3</sup>; Jeremy Wolfe, MD<sup>4</sup>; Eric Chen, MD<sup>5</sup>; Francis C. Decroos, MD<sup>6</sup>; Ehsan Rahimy, MD<sup>7</sup>

<sup>1</sup>The Retina Service of Wills Eye Hospital, Mid Atlantic Retina, Philadelphia, Pennsylvania

### INTRODUCTION

Intravitreal anti-vascular endothelial growth factor (VEGF) agents, including bevacizumab, ranibizumab, and aflibercept, remain the standard of care treatment for neovascular age-related macular degeneration (AMD).<sup>1–4</sup> Various treatment modalities using these agents have been proposed, including monthly, pro re nata, and treat-andextend regimens.<sup>5,6</sup> Despite frequent and consistent treatment with anti-VEGF therapy, there is a subset of patients who are incomplete responders and have persistent exudation, including intraretinal edema, subretinal fluid (SRF), and/or retinal pigment epithelial detachment (PED) on spectral-domain optical coherence tomography (SD-OCT).<sup>7,8</sup>

### **Clinical Data**

While clearance of intravitreal anti-VEGF drugs is not completely understood, some studies have suggested that outflow through the anterior chamber may play a role. 9-12 We hypothesized that by decreasing aqueous production, outflow may also be reduced which could subsequently slow the clearance of intravitreal drugs. In a prior pilot study with 10 eyes of 10 patients who were incomplete responders with neovascular AMD, the effect of topical dorzolamide-timolol in combination with continued intravitreal anti-VEGF injections was explored. Patients were kept on the same anti-VEGF drug as well as the same interval between injections for the 2 visits before enrollment and through the course of the pilot study in order to minimize the chances that any changes noted might be the result of altering one of these variables. The mean central subfield thickness (CST) decreased from 419.7 μm at enrollment to 334.1 μm at the final visit (p=0.012). Mean maximum subretinal fluid (SRF) height decreased from 126.6 μm at enrollment to 56.5

<sup>&</sup>lt;sup>2</sup>Ophthalmic Consultants of Boston, Boston, Massachusetts

<sup>&</sup>lt;sup>3</sup>Tufts Medical Center, Boston, Massachusetts

<sup>&</sup>lt;sup>4</sup>Associated Retinal Consultants at William Beaumont Hospital, Royal Oak, Michigan

<sup>&</sup>lt;sup>5</sup>Retina Consultants of Houston, Houston, Texas

<sup>&</sup>lt;sup>6</sup>Southeastern Retina Associates, Chattanooga, Tennessee

<sup>&</sup>lt;sup>7</sup>Palo Alto Medical Foundation, Palo Alto, California

 $\mu$ m at the final visit (p=0.020). This decrease in mean CST and SRF was significant beginning at the first visit after initiation of the drops.

### **Trial Rationale**

Based on this initial pilot data, dorzolamide-timolol appears to be a promising adjuvant treatment in combination with anti-VEGF injections for incomplete anti-VEGF responders with neovascular AMD. However, since there was no control group in the pilot study, it is possible that the decreased exudation seen was a result of the continued anti-VEGF therapy alone rather than an effect of the topical therapy. As a result, a randomized, placebo-controlled clinical trial will be better able to assess the efficacy of dorzolamide-timolol in this setting.

## TRIAL OBJECTIVES

# **Objective**

The objective of this study is to compare the efficacy of adding topical dorzolamidetimolol versus a topical placebo in combination with intravitreal anti-VEGF injections in patients with neovascular AMD who are anti-VEGF incomplete responders.

## **Endpoints**

# **Primary Efficacy Endpoint:**

The primary efficacy endpoint is change in mean central subfield thickness (CST) on spectral domain optical coherence tomography (SD-OCT) from baseline to the final visit.

# **Secondary Endpoints:**

The secondary endpoints are change in mean maximum subretinal fluid height (SRF), mean maximum pigment epithelial detachment (PED) height, mean intraocular pressure (IOP) and mean pinhole Snellen visual acuity from baseline to final visit.

### TRIAL DESIGN

Subjects will be randomized in a 1:1 ratio to the following groups:

- Topical dorzolamide-timolol 1 drop in study eye twice daily
- Topical artificial tears (placebo group) 1 drop in study eye twice daily

Subjects in both groups will continue to receive the same anti-VEGF drug at the same interval ( $\pm$  1 week) as the 2 visits prior to study enrollment. Once enrolled, subjects will continue on the same drop as initially assigned (dorzolamide-timolol or artificial tears) for the entire study duration starting at baseline and continuing through 3 follow-up visits.

### **PROCEDURES**

## **Vision Testing**

Pinhole Snellen visual acuity will be obtained at each visit.

# **Tonometry**

Tonometry will be performed using either a Tonopen or Goldmann applanation at each visit. If the IOP is  $\geq 25$  mm Hg, Goldmann applanation tonometry must be used to verify the reading.

## **Ophthalmologic Examination**

The following examination will be performed at the baseline visit.

- Inspection of the eyelids
- Examination of the extra-ocular muscle movement
- Inspection of the cornea
- Examination of the anterior chamber for inflammation
- Examination of the pupils
- Examination of the iris
- Inspection of the lens
- Inspection of the vitreous body
- Inspection of the retina and optic disc

# **Optical Coherence Tomography**

Spectral domain optical coherence tomography will be performed at all timepoints. Tracking features should be enabled to allow direct comparison of a given B-scan from one visit to another. In addition, the scan algorithm must allow for automated generation of the central subfield (1 mm circle) thickness.

### SUBJECT POPULATION

## Sample Size

Approximately 50 subjects will be enrolled in the study.

### **Inclusion Criteria**

- 1. Active choroidal neovascularization (CNV) due to AMD.
- 2. Prior treatment with at least 4 injections of anti-VEGF agents in the past 6 months and persistent intraretinal and/or subretinal fluid on SD-OCT at each visit during this period.
- 3. Baseline CST  $\geq$  270  $\mu$ m on SD-OCT automated retinal thickness map.
- 4. Injection of the same anti-VEGF agent (ranibizumab or aflibercept) at each of the two visits immediately preceding study enrollment.
- 5. Time interval of 5 weeks ( $\pm$  1 week) between visits for at least two visits immediately preceding study enrollment.
- 6. Subjects of either gender aged  $\geq$  45 years.

- 7. Provide written informed consent
- 8. Ability to comply with study and follow-up procedures and return for study visits.

### **Exclusion Criteria**

- 1. Anticipated use of intravitreal bevacizumab during the study period
- 2. History of uveitis.
- 3. Presence of intraocular inflammation, significant epiretinal membrane (causing distortion of macular anatomy per investigator discretion), significant vitreomacular traction (per investigator discretion), macular hole, or vitreous hemorrhage.
- 4. Any ophthalmic surgery within previous 6 months, including cataract extraction.
- 5. Any history of vitrectomy or glaucoma surgery (e.g., trabeculectomy, tube shunt).
- 6. Current prescription eye drop usage (e.g., glaucoma drops, corticosteroid drops, etc.).
- 7. Any contraindication for topical use of a beta-blocker (e.g., bradycardia, decompensated heart failure, chronic obstructive pulmonary disease, reactive airway disease, asthma, etc.).
- 8. Any history of sulfonamide allergy.

### TRIAL CONDUCT

Subjects should adhere to the scheduled study visits which will take place at the same interval ( $\pm$  1 week) that they were being injected between the visit prior to enrollment and the enrollment visit (i.e., every 4, 5, or 6 weeks).

### **Overview of Study Assessments**

| Assessment | Baseline | Study Visit 1* | Study Visit 2* | Study Visit 3* |
|---|---|---|---|---|
| Informed Consent | X | | | |
| Medical & | X | | | |
| Ophthalmic History | | | | |
| Vision Testing | X | X | X | X |
| Tonometry | X | X | X | X |
| Ophthalmologic | X | | | |
| Examination | | | | |
| Optical Coherence | X | X | X | X |
| Tomography | | | | |
| Randomization | X | | | |
| Subjects Randomized | | | | |
| to DorzolamideTimolol | | | | |
| Reminded to | X | X | X | |
| Use Drops and Given | | | | |
| Bottle | | | | |

| Bottle |
|--------|
|--------|

<sup>\*</sup>Interval between each visit will be based upon the interval between the visit prior to enrollment and the enrollment visit. Subjects should be encouraged to follow-up at this same interval (± 1 week) for the duration of the study.

# **Study Assessments**

The following evaluations will be performed at the visits specified below.

## Baseline (Day of Enrollment in Study)

## **Pre-injection**

- Vision testing
- Ophthalmologic examination and tonometry
- Optical coherence tomography

# **Injection**

- Optional if patient consents separately: Aqueous humor sample prior to antiVEGF injection
- Intravitreal injection of same anti-VEGF drug used at the two visits prior to enrollment (i.e., ranibizumab or aflibercept).

## Post-injection

• Instruct patient on use of topical drop (dorzolamide-timolol vs. artificial tears as assigned at randomization, 1 drop twice daily for study duration) to begin same day.

## Study Visit 1

## Pre-injection

- Vision testing and tonometry
- Optical coherence tomography

## **Injection**

- Optional if patient consents separately: Aqueous humor sample prior to antiVEGF injection
- Intravitreal injection of same anti-VEGF drug used previously (i.e., ranibizumab or aflibercept ).

### Post-injection

• Instruct patient on continuing use of topical drop (dorzolamide-timolol vs. artificial tears as previously assigned, 1 drop twice daily for study duration) to begin same day.

## Study Visit 2

### Pre-injection

- Vision testing and tonometry
- Optical coherence tomography

## **Injection**

• Intravitreal injection of same anti-VEGF drug used previously (i.e., ranibizumab or aflibercept).

## Post-injection

• Instruct patient on continuing use of topical drop (dorzolamide-timolol vs. artificial tears as previously assigned, 1 drop twice daily for study duration) to begin same day.

## Study Visit 3

### Pre-injection

- Vision testing
- Ophthalmologic examination and tonometry
- Optical coherence tomography

## **Aqueous Humor Samples (optional)**

Anterior chamber (aqueous humor) samples will be collected from all patients who provide additional consent to participate. Where patient consents to aqueous humor sampling, all efforts should be made to collect a baseline aqueous humor sample on the Baseline visit and Study Visit 1.

#### Withdrawal from Trial

Subjects have the right to withdraw from the trial at any time for any reason. The investigator also has the right to withdraw subjects from the trial in the event of concurrent illness, adverse events, treatment failure after a prescribed procedure, protocol violations, cure, administrative or other reasons.

## STATISTICAL METHODS

## **Experimental Design**

This is a randomized clinical trial in which 50 subjects will be randomly assigned to receive topical dorzolamide-timolol or artificial tears (1 drop twice daily for the study duration) in combination with continuing intravitreal anti-VEGF injections for neovascular AMD.

## **Sample Size**

Assuming a power of 0.9 and an alpha of 0.05, approximately 44 patients will be required to demonstrate a CST improvement of 400 to 350 microns with a standard deviation of 50 microns. Estimating a 10% drop out rate, approximately 50 patients will be targeted for enrollment.

### Statistical Analysis (finalized 2/4/20)

Statistical analyses were not pre-specified. Snellen VA was converted to logMAR for analysis. For continuous variables, the mean difference and 95% confidence intervals

between the two groups were derived using analysis of covariance (ANCOVA) with the baseline value and type of anti-VEGF drug used as covariates. For binary outcomes, a logistic regression was used with the baseline value as a covariate. Missing data were excluded from analyses such that complete-case analysis was conducted and multiple secondary outcomes were evaluated without formal control for multiplicity, i.e., without adjustment for multiple analyses. All *P* values were two-sided. A *P* value < .05 was considered statistically significant for the primary outcome, and a *P* value < .001 was considered statistically significant for any other outcomes since there was no adjustment for multiple analyses.

## References

- 1. Moshfeghi AA, Rosenfeld PJ, Puliafito CA, et al. Systemic bevacizumab (Avastin) therapy for neovascular age-related macular degeneration: twenty-four-week results of an uncontrolled open-label clinical study. Ophthalmology 2006;113:2002.e1–12.
- 2. Rosenfeld PJ, Brown DM, Heier JS, et al. Ranibizumab for neovascular agerelated macular degeneration. N Engl J Med 2006;355:1419–1431.
- 3. Heier JS, Brown DM, Chong V, et al. Intravitreal aflibercept (VEGF trap-eye) in wet age-related macular degeneration. Ophthalmology 2012;119:2537–2548.
- 4. Bressler NM. Antiangiogenic approaches to age-related macular degeneration today. Ophthalmology 2009;116:S15–23.
- 5. Brown DM, Regillo CD. Anti-VEGF agents in the treatment of neovascular agerelated macular degeneration: applying clinical trial results to the treatment of everyday patients. Am J Ophthalmol 2007;144:627–637.
- 6. Arnold JJ, Campain A, Barthelmes D, et al. Two-year outcomes of "treat and extend" intravitreal therapy for neovascular age-related macular degeneration. Ophthalmology 2015;122:1212–1219.
- 7. Krebs I, Glittenberg C, Ansari-Shahrezaei S, et al. Non-responders to treatment with antagonists of vascular endothelial growth factor in age-related macular degeneration. Br J Ophthalmol 2013;97:1443–1446.
- 8. Barthelmes D, Walton R, Campain AE, et al. Outcomes of persistently active neovascular age-related macular degeneration treated with VEGF inhibitors: observational study data. Br J Ophthalmol 2015;99:359–364.
- 9. Byeon SH, Kwon OW, Song JH, et al. Prolongation of activity of single intravitreal bevacizumab by adjuvant topical aqueous depressant (Timolol-Dorzolamide). Graefes Arch Clin Exp Ophthalmol 2009;247:35–42.
- 10. Bakri SJ, Snyder MR, Reid JM, et al. Pharmacokinetics of intravitreal bevacizumab (Avastin). Ophthalmology 2007;114:855–859.
- 11. Stewart MW. Predicted biologic activity of intravitreal bevacizumab. Retina 2007;27:1196–1200.
- 12. Gaudreault J, Fei D, Rusit J, et al. Preclinical pharmacokinetics of Ranibizumab (rhuFabV2) after a single intravitreal administration. Invest Ophthalmol Vis Sci 2005;46:726–733.

13. Sridhar J, Hsu J, Shahlaee A, Garg SJ, Spirn MJ, Fineman MS, Vander J. Topical dorzolamide-timolol with intravitreous anti-vascular endothelial growth factor for neovascular age-related macular degeneration. JAMA Ophthalmol 2016 Feb 25. doi: 10.1001/jamaophthalmol.2016.0045